CLINICAL TRIAL: NCT04753164
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Proof-of-concept Study to Evaluate the Efficacy and Safety of Oral ACT-539313 in the Treatment of Adults With Moderate to Severe Binge Eating Disorder
Brief Title: Multicenter Study to Evaluate the Efficacy and Safety of Oral ACT-539313 in the Treatment of Adults With Moderate to Severe Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-082A201
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — ACT-539313

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled, parallel-group, proof-of-concept study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg twice daily (b.i.d.) ACT-539313 (Experimental)
  Interventions: Drug: ACT-539313
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-539313 — ACT-539313 as capsules at a strength of 100 mg, taken orally, b.i.d. in the morning at breakfast and in the evening at dinner, with a glass of water during the treatment period.
  Arms: 100 mg twice daily (b.i.d.) ACT-539313
Drug: Placebo — Matching placebo as identical capsules indistinguishable from ACT-539313, taken orally, b.i.d. in the morning at breakfast and in the evening at dinner, with a glass of water during the treatment period.
  Arms: Placebo

SUMMARY:
Placebo-controlled study to evaluate the efficacy and safety of oral ACT-539313 in the treatment of adults with moderate to severe binge eating disorder

ELIGIBILITY:
Inclusion Criteria:

Criteria assessed at Visit 1:

* Signed and dated informed consent form prior to any study-mandated procedure.
* Male or female study participants aged 18 to 55 years at the time of signing the informed consent form.
* Binge-eating disorder (BED) in accordance with Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria diagnosed using the Structured Clinical Interview for DSM-5 (SCID-5).
* Self-reported BED severity of at least moderate level, defined as at least 4 BE episodes per week, on average, for a duration of at least 6 months.
* BED in accordance with Eating Disorder Examination Questionnaire (EDE-Q).
* Clinical Global Impression of Severity scale (CGI-S) score of ≥ 4.
* For women of childbearing potential (WOCBP): Negative serum pregnancy test at Visit 1; agreement to undertake monthly urine or serum pregnancy tests during the study and up to the EOS visit; agreement to use an acceptable contraceptive method.

Criteria assessed at Visit 2:

* Reporting ≥3 BE days for each of the 2 weeks prior to randomization as documented in the participant's BE diary and with BE diary entries completed for at least 6 days per week during this 2-week period (between Visit 1 and 2).
* CGI-S score of ≥ 4.
* For WOCBP: negative urine pregnancy test.

Exclusion Criteria:

Criteria assessed at Visit 1:

* BMI < 18.0 kg/m² or > 45 kg/m².
* Any acute or chronic-persistent psychiatric disorder other than BED diagnosed in the past, including anorexia nervosa, bulimia, psychotic disorders, bipolar disorder, hypomania, or dementia, as defined by the DSM-5 criteria or by the Mini International Neuropsychiatric Interview (MINI©).
* Use of any medications for the treatment of BED (including lisdexamfetamine [Vyvanse®]), any other eating disorder, obesity, or weight gain, or any other medication that could result in weight gain or weight loss, including over-the-counter and herbal products, within 3 months prior to Screening.
* Any clinically unstable medical condition, significant medical disorder or acute illness that, in the investigator's opinion, could interfere with the participants ability to comply with study assessments or abide by study restrictions.

Criteria assessed at Visit 1 and Visit 2

* HAMD-17 score ≥ 17 points at Visit 1 and/or Visit 2.
* Any of the following conditions related to suicidality:

  1. Participant is considered to have a suicide risk in the investigator's opinion or has a previous history of suicide attempt within the past 12 months.
  2. Participant answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS© assessment at Screening (in the past month). Participants who answer "yes" to this question must be referred to the investigator for follow-up evaluation.
* Female participants: pregnant, lactating or planning to become pregnant during the projected course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (30):
- United States (30):
  - Southern California Research, Beverly Hills, California
  - Wr-Pri, Llc, Encino, California
  - Collaborative Neuroscience Network (CNS), Garden Grove, California
  - Syrentis Clinical Research, Santa Ana, California
  - Connecticut Clinical Research - Cromwell, Cromwell, Connecticut
  - Clinical Neurosciences Solutions, Jacksonville, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - NeuorTrials Research Inc, Atlanta, Georgia
  - Psych Atlanta P.C., Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Collective Medical Research, Prairie Village, Kansas
  - Harvard Medical School - McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Inc, Boston, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - St. Charles Psychiatric Associates dba Midwest research group, Saint Charles, Missouri
  - M3 Wake Research, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - Bioscience Research, Mount Kisco, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - The Medical Research Network, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - University of Cincinnati College of Medicine - Lindner Center of HOPE, Mason, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center For Clinical Inv., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 sites in the USA; all 26 sites randomized subjects.
Pre-assignment Details: In total, 259 subjects were screened, of which 123 discontinued during the screening period.
Period: Overall Study
Arm/Group | 100 mg Twice Daily (b.i.d.) ACT-539313 | Placebo
Started | 68 | 68
Completed | 41 | 48
Not Completed | 27 | 20
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Lost to Follow-up | 6 | 6
Not completed — Other | 12 | 5

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Twice Daily (b.i.d.) ACT-539313 | Placebo | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Median (Full Range); unit: years] — Population: Randomized population
  years | 37 [20 to 55] | 42 [18 to 55] | 39 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomized population
  Participants
    Female | 55 | 50 | 105
    Male | 13 | 18 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Randomized population
  Participants
    Hispanic or Latino | 14 | 16 | 30
    Not Hispanic or Latino | 53 | 51 | 104
    Unknown or Not Reported | 1 | 1 | 2
Body mass index (kg/m^2) at screening [Mean (Standard Deviation); unit: kg/m2] — Population: Randomized population; Number analyzed in the "Placebo" group n = 67; missing: n = 1
  kg/m2
    number analyzed (Participants) | 68 | 67 | 135
    (all) | 35.03 (6.99) | 34.93 (6.01) | 34.98 (6.50)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Number of Binge Eating (BE) Days Per Week
Description: BE days per week is defined as the number of diary days with at least one confirmed BE episode during the applicable 14-day time interval divided by the total number of diary days, times 7.
Time Frame: From baseline to Week 12; duration approx. 3.5 months
Population: Full Analysis Set; subjects with available data for calculation of the change from baseline at Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: BE days per week
Arm/Group | 100 mg Twice Daily (b.i.d.) ACT-539313 | Placebo
Number analyzed (Participants) | 43 | 45
BE days per week | -2.93 [-3.46 to -2.40] | -2.93 [-3.47 to -2.39]
Statistical Analysis 1: Comparison: 100 mg Twice Daily (b.i.d.) ACT-539313 vs Placebo; Test type: Other — Mixed effects model for Repeated Measures: Change from baseline in the number of BE days per week = baseline number of BE days per week + sex (Male; Female) + BMI group (< 30 ; ≥ 30 kg/m2) + treatment + visit + treatment × visit + baseline × visit; p = 0.9992, Mixed effects model f. repeated measures; LS Mean Difference to Placebo = 0.00, 95% CI 2-sided [-0.69 to 0.69]

ADVERSE EVENTS:
Time Frame: AEs reported are AEs occurring or worsening during the treatment period; duration approx. 3 months.
Arm/Group | 100 mg Twice Daily (b.i.d.) ACT-539313 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/68
Other Adverse Events (participants affected / at risk) | 31/68 | 25/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Twice Daily (b.i.d.) ACT-539313 (N=68) | Placebo (N=68)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Twice Daily (b.i.d.) ACT-539313 (N=68) | Placebo (N=68)
Somnolence (Nervous system disorders) | 9 | 13
Accidental overdose (Injury, poisoning and procedural complications) | 8 | 7
Fatigue (General disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 5 | 1
Headache (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04753164/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT04753164/SAP_001.pdf